CLINICAL TRIAL: NCT02462902
Title: Comparison And Outcomes Of Fluid Resucitation With 0.9% Normal Saline And 5% Albumin In Cirrhosis Patients With Sepsis Induced Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis with sepsis-01
Record Dates: First submitted 2015-05-25; First posted 2015-06-04 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-05

CONDITIONS: Cirrhosis With Septic Shock
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5% albumin Infusion (Experimental): (250 ml over 15 to 30 minutes)
  Interventions: Drug: 5% albumin Infusion
- 0.9% sodium chloride solution (Active Comparator): 0.9% sodium chloride solution (total of 30ml/kg over 15 to 30 minute)
  Interventions: Drug: 0.9% sodium chloride solution

INTERVENTIONS:
Drug: 5% albumin Infusion — colloid, 5% albumin (250 ml over 15 to 30 minutes).
  Arms: 5% albumin Infusion
Drug: 0.9% sodium chloride solution — 0.9% sodium chloride solution (total of 30ml/kg over 15 to 30 minutes)
  Arms: 0.9% sodium chloride solution

SUMMARY:
300 consecutive patients with cirrhosis of any aetiology admitted with features of sepsis and sepsis induced hypotension to the intensive care unit, the emergency department and the step down units of Institute of Liver and Biliary Sciences, New Delhi, who fulfil the inclusion criteria.

This study will be a single centre prospective randomized comparative trial. Patients will be randomized into two groups. Group A will receive crystalloid, 0.9% sodium chloride solution (total of 30ml/kg over 30 minutes) and Group B will receive colloid, 5% albumin (250 ml over 15 minutes).

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhotic patients of any aetiology with Infection - suspected or documented and Mean arterial pressure less than 65 mm of Hg

Exclusion Criteria:

1. Cirrhosis patients in septic shock who are already on vasopressors and/or inotropes
2. Cirrhosis patients in septic shock with structural heart disease
3. Cirrhosis patients in septic shock with chronic renal failure/dialysis dependent/volume overloaded state
4. Cirrhosis patients in shock, caused by other reasons, other than septic shock
5. Cirrhosis patients in septic shock in whom contraindication to internal jugular or subclavian line insertion is present
6. Age less than 18 years
7. Previous episode of septic shock during the same hospital stay
8. Pregnant or lactating women
9. Patients in need for emergent surgical interventions
10. Cirrhosis patients in septic shock with chronic obstructive lung disease and right heart failure
11. Cirrhosis patients in septic shock with associated upper gastrointestinal bleed or coagulopathy related bleed with a haemoglobin of less than 8g/dL or requiring urgent transfusions of blood and blood products
12. A previous adverse reaction to human albumin solution

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Total number of patients with MAP (Mean Arterial Pressure) ≥ 65 | 3 hours

SECONDARY OUTCOMES:
Change in lactate dynamics | 3 hours
Total number of patients with Urine output >/= 0.5mL/kg/hr. | 3 hours
Mortality | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India